CLINICAL TRIAL: NCT02232932
Title: Randomized Prospective Multicentric Study: Radio-chemotherapy and Liver Transplantation Versus Liver Resection to Treat Respectable Hilar Cholangiocarcinoma
Brief Title: Liver Resection Versus Radio-chemotherapy-Transplantation for Hilar Cholangiocarcinoma
Acronym: TRANSPHIL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120106
Record Dates: First submitted 2014-08-06; First posted 2014-09-05 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Cholangiocarcinoma
Keywords: Hilar cholangiocarcinoma; Liver transplantation; Radiochemotherapy
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor | interventions — Liver Transplantation; Hepatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CAPECITABINE-Radiotherapy -Liver Transplantation (Experimental): Neoadjuvant Radio-Chemotherapy (RC) and Liver Transplantation (LT)
  Interventions: Procedure: CAPECITABINE-Radiotherapy -Liver Transplantation
- RESECTION (Active Comparator): Liver resection
  Interventions: Procedure: RESECTION

INTERVENTIONS:
Procedure: CAPECITABINE-Radiotherapy -Liver Transplantation — CAPECITABINE (800 mg/m2 twice a day during 5 weeks) + External Radiotherapy (50 grays during 5 weeks) then Liver transplantation
  Other Names: Neoadjuvant Radio-Chemotherapy and Liver Transplantation
  Arms: CAPECITABINE-Radiotherapy -Liver Transplantation
Procedure: RESECTION — Intent-to-treat R0 liver resection
  Other Names: Liver Resection
  Arms: RESECTION

SUMMARY:
A prospective, open-label, randomised, multicentre, comparative study in two parallel groups comparing an interventional group with liver transplantation preceded by neoadjuvant radio-chemotherapy and a control group receiving conventional liver and bile duct resection.

The primary endpoint will be overall survival at 5 years in the intent-to-treat population. The secondary endpoint will be recurrence-free survival at 3 years evaluated by CT-scan and tumoral markers (Carcinoembryonic antigen (CAE) and cancer antigen (CA19.9)) in the intent-to-treat population.

The number of subjects necessary is 54 patients (27 x 2): this population will enable the demonstration of a significant difference is 5-year survival rates between the transplanted group and the resected group with a power of 80% and a first-species risk of 5%, under the hypothesis that these survival rates are 70% in the transplanted group and 30% in the resected group.

DETAILED DESCRIPTION:
The protocol will comprise a phase 1 during which the potential eligibility of patients (presenting with a resectable Klatskin - Excepted Type 1of Bismuth) will be assessed, based on clinical, biological and morphological data. After phases 1, the eligibility of the patient will be confirmed or not. In the context of the study, phase 2 will include the collection of blood samples as well as positon emission tomography (PET)-scan and upper endoscopic ultrasound (EUS) in order to rule out any obvious lymph node metastases. A short exploratory laparoscopy will also be performed in phase 2 to eliminate infra-clinic subcapsular liver metastases and peritoneal carcinomatosis. The randomization process will take place at the end of the phase 2, patients will be assigned into the transplantation arm (OLT) or the resection arm (RSX). During phase 3, patient will receive nutritional support and, if not done previously, a biliary drainage will be placed endoscopically. In the RSX arm (phase 3A), patients will undergo radical resection of the tumor (refer below technical details). Preoperative portal vein embolization may be necessary at this stage depending on the expected remnant liver volume, assessed by CT-scan volumetry. In the OLT arm (phase 3A), patients will receive neoadjuvant radiochemotherapy (External - 50 grays) following by liver transplantation (phase 4B). Before the fifth week after completion of radiochemotherapy, a staging laparotomy with local lymphadenectomy will be performed and patients will be put on the national waiting list in the absence of extra-hepatic disease, especially peritoneal seeding and lymph nodes involvement. A score exception will allowed a liver transplantation in the 3 months after staging laparotomy. During phase 5 the patient will be monitored postoperatively at the clinical, biological and morphological levels for 3 months. During phase 6, the patient will be followed clinically, biologically and morphologically for 5 years in order to detect any recurrence and in the context of standard clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male or female) aged from 18 to 68 year-old, French
* Hilar cholangiocarcinoma histologically proved and/or highly suspected on hilar stenosis with mass syndrome from 0.1 cm to 3 cm
* Hilar cholangiocarcinoma type 2, type 3A, type 3B, type 4
* Patients considered as resectable (R0 resection) by liver resection including segment 1 and biliary confluence with or without vascular resection
* Patient potentially transplantable
* Patient affiliated to French Health Insurance
* Patient who had sign an informed consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Women of childbearing potential without an effective contraception method
* Radiotherapy contraindication
* Positive dosage of ImmunoglobulinsG4 (IgG4)
* dihydro-pyrimidine-dehydrogenase (DPD) total deficit
* Personal history of cancer in the last 5 five years (exclusion basocellular cellular carcinoma)
* Personal history of fluoropyrimidine hypersensibility
* Personal history of capecitabine hypersensibility
* Personal history of dihydro-pyrimidine-dehydrogenase deficit
* Polynuclear neutrophil < 1500 / ml
* Platelet rate < 100 000 / ml
* Severe leucopenia < 2000 / ml
* Severe liver failure (Factor V < 50%)
* Severe renal failure (Creatin clearance < 30 ml/min)
* Treatment by Sorivudine or its analogue as Brivudine
* Non controled diabetes mellitus and/or others severe co-morbidities (renal failure, severe and instable coronaropathy, severe risk factor of stroke, body mass index superior to 35)
* Proved histological cirrhosis
* Sclerosing cholangitis
* Intra and/or extra-hepatic metastases
* Hypereosinophilia and/or wirsung dilatation and/or mass of the pancreas head
* Hilar mass superior to 3 cm
* Duodenal invasion
* Patient under guardianship

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-02 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At 5 years
  To demonstrate the superiority, in terms of 5-year survival, of liver transplantation (TH) preceded by neoadjuvant chemoradiotherapy on the radical resection of Klatskin tumors considered resectable

SECONDARY OUTCOMES:
Recurrence free survival | At 3 years
  3-year recurrence-free survival assessed by CT and markers

CONTACTS AND LOCATIONS:
Overall Officials: Eric VIBERT, MD, Principal Investigator — AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif, France
Locations (1):
- AP-HP, Paul Brousse Hospital, Centre Hepato-Biliaire, Villejuif, France